CLINICAL TRIAL: NCT02201693
Title: Randomised Trial Comparing 12 Months of Cyclic Enteral Nutrition to Supplementary Enteral Nutrition as Maintenance Therapy for Pediatric Crohn's Disease
Brief Title: Cyclic Exclusive Enteral Nutrition as Maintenance Therapy for Pediatric Crohn's Disease
Acronym: CD-HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GETAID Pediatric (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130302; 2013-A01473-42 (Other: ANSM)
Record Dates: First submitted 2014-07-17; First posted 2014-07-28 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease,; pediatric GETAID (Therapeutic study group of inflammatory bowel diseases of the child),; enteral nutrition,; randomized multicenter study
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclic exclusive MODULEN IBD (Experimental): Cyclic exclusive MODULEN IBD for 2 weeks every 8 weeks
  Interventions: Dietary Supplement: MODULEN IBD
- MODULEN IBD supplementation (25% of caloric requirements) (Experimental): MODULEN IBD supplementation (25% of caloric requirements) alone A Physician not involved in the study design and blinded to the treatment arm will perform the evaluation of the patients during each study visit.
  Interventions: Dietary Supplement: MODULEN IBD

INTERVENTIONS:
Dietary Supplement: MODULEN IBD — 2 week ON / 6 weeks OFF treatment every 8 weeks covering at least 100% of daily caloric requirement (approx. 2-2.5L/day).
  Arms: Cyclic exclusive MODULEN IBD
Dietary Supplement: MODULEN IBD — 25% of daily caloric requirements, approx. 500mL/day
  Arms: MODULEN IBD supplementation (25% of caloric requirements)

SUMMARY:
The purpose of this study is to compare the rate of first relapse at 12 months between maintenance therapy with cyclic exclusive enteral nutrition (EEN) (at least 100% daily calories) and maintenance therapy with supplementary enteral nutritional support (25% daily calories).

DETAILED DESCRIPTION:
Enteral nutrition (EN) is a highly efficacious treatment option for Crohn's disease (CD). In children, exclusive EN is considered first choice therapy to induce remission in pediatric CD, as highlighted in the recent ESPGHAN-ECCO guidelines. Several meta-analyses showed that the anti-inflammatory potential of EEN is comparable to the effects of steroids. In addition, children with CD often have marked growth retardation and EEN is one of the most efficacious treatment options to induce catch-up growth in these patients. There is convincing data indicating that EN is highly efficacious when given on an exclusive basis, while the use of partial EN is markedly less effective to induce remission in active Crohn's disease as compared to exclusive EN. Recently, it was suggested that exclusive EN has a dominant effect on the intestinal microbiota, which contributes to the induction of remission. There exists several strategies to maintain remission in children with CD, but there is no clear consensus on which maintenance treatment to follow. There are some indicators to believe that enteral nutritional therapy might play also a significant role as maintenance therapy for CD. Given the fact that many centers use a top-down approach with the introduction of immunosuppressors and/or biologics at/or shortly after diagnosis, the investigators wanted to test the possibility of a treatment option to efficiently maintain remission with less (or no) side effects based on enteral nutrition to avoid the early use of immunosuppressors.

It's a French multicenter, prospective, randomized study with PROBE (prospective randomized open blind end-point) evaluation. Randomization will be performed in a blinded and centralized manner, allocating patients to one of the two treatment groups :

* ARM A : Cyclic exclusive MODULEN IBD for 2 weeks every 8 weeks
* ARM B: MODULEN IBD supplementation (25% of caloric requirements) alone

A Physician not involved in the study design and blinded to the treatment arm will perform the evaluation of the patients during each study visit.

A total of four visits (including final visit) are scheduled for this trial over a period of 12 months at a rhythm of every three months (+/- 2 weeks) for all patients. The study visit will happen during scheduled routine visits, necessary for the routine care of CD patients. Each visit comprises a routine clinical evaluation. The assessment of maintenance of remission is particularly important (wPCDAI<12.5 points), a routine lab analysis including fecal calprotectin is required at each visit. In addition, all relevant medical or other events will be recorded. Only for patients who participate in the annex studies an additional stool sample (microbial analysis) is required. At M9 visit, follow-up endoscopy (M12+/- 6weeks) and entero-MRI (M12+/- 6 weeks) will be programmed as part of the routine surveillance of patients on maintenance therapy, allowing to adjust treatment in the following if necessary. Compliance to treatment will be monitored by recordings of daily MODULEN IBD intake during 2 week periods on the E-system. A quality of life E-questionnaire will be filled out one day prior to each visit.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years
* Confirmed Crohn's disease (L1, L2, L3+/- L4a/b)
* new-onset disease or acute relapse treated with enteral nutrition
* responding to induction therapy with exclusive enteral nutrition with complete clinical remission at inclusion visit (wPCDAI<12.5)
* completed cycle of induction therapy of at least 6 weeks (6-12 weeks)
* biological treatment by Remicade has to be stopped at least 8 weeks prior to inclusion
* "wash out" of corticosteroids, immunosuppressors and treatment by Humira of minimally 4 weeks prior to inclusion
* 5-ASA and derivates have to be stopped at least at screening visit
* Antibiotics must be stopped at least 2 weeks prior to inclusion
* Informed and signed consent

Exclusion Criteria:

* Patients with B2 or B3 disease behavior (intestinal/colonic stenosis (including ileo-caecal valve), intrabdominal abscess, fistulizing disease)
* Patients not in remission on induction therapy (wPCDAI>12.5)
* Patients with isolated and severe perianal disease
* Patients requiring surgical therapy at inclusion
* Ongoing steroid medication
* Ongoing immunosuppressor or biologics therapy
* No informed consent
* Currently participating or having participated in another interventional clinical trial during the last 4 weeks prior to the beginning of this study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
The first relapse | 12 months
  Assessed with wPCDAI

SECONDARY OUTCOMES:
Clinical remission | 12 months
  Assessed with wPCDAI, CDAI, PGA
Time to the first relapse | until month 12
  Assessed with wPCDAI, CDAI, PGA
Variation of wPCDAI, | until month12
  Assessed with wPCDAI
Endoscopic remission | month 12
  CDEIS
Transmural healing | Month 12
  MRI
Calprotectin | until month12
  Fecal sample
Quality of life analysis | Until Month 12
  E-questionnaire
Growth pattern | Until Month 12
  Z-Score

CONTACTS AND LOCATIONS:
Overall Officials: Franck RUEMMELE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker - Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pigneur B, Martinez-Vinson C, Bourmaud A, Dabadie A, Duclaux-Loras R, Hugot JP, Roman C, Dumant C, Spyckerelle C, Guinard-Samuel V, Willot S, Dupont C, Breton A, Caron N, Chaillou E, Rebouissoux L, Bertrand V, Triolo V, Pages J, Djeddi D, Bonneton M, Uhlen S, Catteau N, Coopman S, Lepage P, Viala J, Ruemmele FM. Cyclic exclusive enteral nutrition versus partial enteral nutrition to maintain long-term drug-free remission in paediatric Crohn's disease (CD-HOPE): an open-label, endpoint-blinded, randomised controlled trial. Lancet Gastroenterol Hepatol. 2026 Jan 19:S2468-1253(25)00262-6. doi: 10.1016/S2468-1253(25)00262-6. Online ahead of print. PMID 41570843